CLINICAL TRIAL: NCT04162899
Title: A Randomized, Double-Blind and Placebo-Controlled Phase II Study to Evaluate the Efficacy and Safety of SHR0302 in Adult Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Phase II Study in Adult Patients With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSJ10303
Record Dates: First submitted 2019-10-15; First posted 2019-11-14 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — ivarmacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Comparator: SHR0302 dose A (Active Comparator): Participants randomized in this arm will receive dose A of SHR0302 until end of study at week 12.
  Interventions: Drug: Drug: SHR0302
- Active Comparator: SHR0302 dose B (Active Comparator): Participants randomized in this arm will receive dose B of SHR0302 until end of study at week 12.
  Interventions: Drug: Drug: SHR0302
- Placebo Comparator: Placebo (Active Comparator): Participants randomized in this arm will receive Placebo of SHR0302 until end of study at week 12.
  Interventions: Drug: Drug: SHR0302

INTERVENTIONS:
Drug: Drug: SHR0302 — The study drug, SHR0302, is designed to block the activity of an enzyme protein called JAK-1(known as a JAK-1 inhibitor).

SUMMARY:
This proposed study is a randomized, double-blind, placebo-controlled, 3-arm parallel, multicenter phase II study, designed to explore the efficacy and safety of SHR0302 treatment for patients with moderate to severe atopic dermatitis.

The study will be conducted over a 12-week treatment period. Two active doses of SHR0302 will be compared to placebo and improvement in atopic dermatitis will be assessed using the Investigator's Global Score (IGA)

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18-75 years of age (inclusive), male or female, at the time of informed consent
* Moderate to severe atopic dermatitis
* Capable of providing a signed and dated informed consent form indicating the subject has been informed of all pertinent aspect of the study

Exclusion Criteria:

* Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study
* Subject has a current diagnosis of other active skin disease (e.g., psoriasis or lupus erythematosus) or skin infection (bacterial, fungal, or viral) that may affect the evaluation of atopic dermatitis
* Subject has a severe comorbidity that may require systemic steroids therapy or other interventions or requires active frequent monitoring (e.g., unstable chronic asthma)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - Peking University People's Hospital, Xicheng, Beijing Municipality
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - Xuanwu Hospital Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Peking union medical college hospital, Beijing
  - Beijing Tsinghua Changgeng Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital of Central South University, Changsha
  - The Third Xiangya Hospital of Central South University, Changsha
  - Second Affiliated Hospital of Army Medical University (Xinqiao Hospital), Chongqing
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun. Yat- Sen Memorial Hospital, Sun. Yat- Sen University, Guangzhou
  - The first affiliated hospital Zhejiang university, Hangzhou
  - Affiliated Hangzhou first people's hospital, Zhejiang university school of medicine, Hangzhou
  - Zhejiang province People's Hospital, Hangzhou
  - Jinan Central Hospital, Jinan
  - Shanghai Skin Disease Hospital, Shanghai
  - The first hospital of China medical university, Shenyang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - The First Hospital of Shanxi Medical University, Taiyuan
  - Union Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Henan provincial people's hospital, Zhengzhou

REFERENCES:
- [Derived] Zhao Y, Zhang L, Ding Y, Tao X, Ji C, Dong X, Lu J, Wu L, Wang R, Lu Q, Goh AH, Liu R, Zhang Z, Zhang J. Efficacy and Safety of SHR0302, a Highly Selective Janus Kinase 1 Inhibitor, in Patients with Moderate to Severe Atopic Dermatitis: A Phase II Randomized Clinical Trial. Am J Clin Dermatol. 2021 Nov;22(6):877-889. doi: 10.1007/s40257-021-00627-2. Epub 2021 Aug 9. PMID 34374027

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Comparator: SHR0302 Dose A | Active Comparator: SHR0302 Dose B | Placebo Comparator: Placebo
Started | 35 | 35 | 35
Completed | 29 | 32 | 23
Not Completed | 6 | 3 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: SHR0302 Dose A | Active Comparator: SHR0302 Dose B | Placebo Comparator: Placebo | Total
Number analyzed (Participants) | 35 | 35 | 35 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (14.79) | 35.2 (14.75) | 30.3 (12.59) | 34.7 (14.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 9 | 36
  Male | 20 | 23 | 26 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 35 | 35 | 105
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 35 | 35 | 35 | 105
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Disease duration [Mean (Standard Deviation); unit: years] | 10.91 (10.214) | 8.95 (8.468) | 8.67 (7.624) | 9.51 (8.807)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Achieving Investigator's Global Assessment (IGA) Response Which Improvement ≥ 2 From Baseline.
Description: The IGA is a validated assessment instrument used in clinical studies to rate the severity of AD globally. IGA response was defined as IGA score of 0/1 (complete or almost complete clearance of skin lesions) with an improvement in IGA score by ≥ 2 from baseline.
Time Frame: At week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator: SHR0302 Dose A | Active Comparator: SHR0302 Dose B | Placebo Comparator: Placebo
Number analyzed (Participants) | 35 | 35 | 35
Participants | 9 | 19 | 2

2. Secondary Outcome: Percentage of Czema Area and Severity Index (EASI) Change.
Description: The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of atopic dermatitis (AD).
Time Frame: Up to week 12
Reporting Status: Not Posted

3. Secondary Outcome: Percentage of Subjects Achieving Investigator's Global Score (IGA) Response
Description: The IGA is a validated assessment instrument used in clinical studies to rate The IGA is a validated assessment instrument used in clinical studies to rate the severity of AD globally.
Time Frame: Up to week 8
Reporting Status: Not Posted

4. Secondary Outcome: Percent of Pruritus Numerical Rating Scale (NRS) Change
Description: The Pruritus NRS is an assessment tool that participants used to report the intensity of their pruritus during a 24-hour recall period.
Time Frame: Up to week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Active Comparator: SHR0302 Dose A | Active Comparator: SHR0302 Dose B | Placebo Comparator: Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 2/35 | 1/35 | 0/35
Other Adverse Events (participants affected / at risk) | 13/35 | 16/35 | 10/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator: SHR0302 Dose A (N=35) | Active Comparator: SHR0302 Dose B (N=35) | Placebo Comparator: Placebo (N=35)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator: SHR0302 Dose A (N=35) | Active Comparator: SHR0302 Dose B (N=35) | Placebo Comparator: Placebo (N=35)
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 0
Blood pressure increased (Investigations) | 0 | 2 | 0
Transaminases increased (Investigations) | 2 | 1 | 3
Tri-iodothyronine free increased (Investigations) | 2 | 1 | 4
Weight decreased (Investigations) | 0 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Headache (Nervous system disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT04162899/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT04162899/SAP_001.pdf